CLINICAL TRIAL: NCT05934279
Title: Developing an Effective Intervention to Address Post-COVID-19 Balance Disorders, Weakness and Muscle Fatigue in Individuals Aged 65+
Brief Title: Developing an Effective Intervention to Address Post-Corona-Virus-Disease-2019 Balance Disorders, Weakness and Muscle Fatigue in Individuals Aged 65+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKE 01-41/2022
Record Dates: First submitted 2023-01-03; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: post-COVID-19; elderly individuals; balance disorder
MeSH Terms: conditions — COVID-19 | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The participants will be randomized to one of 2 groups: RT and control (no exercise). The participants' muscle strength under dynamic condition, balance (especially fall risk), body composition and quality of life will be assessed pre- and post-intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training (Experimental): Training aimed at improving balance and strengthening muscle strength (RT) will be held twice a week, 45 min per session for 8 weeks
  Interventions: Device: Resistance Training
- Control Group (No Intervention): Group without training program

INTERVENTIONS:
Device: Resistance Training — All training exercise involve balance and strength improvement. Consist of 8 weeks of trainings per 2 trainings in each week, ongoing 45 minutes.
  Arms: Resistance Training

SUMMARY:
The long-term consequences and sequelae of COVID-19 are still unclear; however, a vast number of elderly individuals have reported prolonged general weakness and muscular fatigue, leading to significant functional decline, increased risk of falls, morbidity and mortality rates. However, effective exercise intervention for such post-COVID-19 patients is still not well documented. Previous studies indicate that, in general, resistance training (RT) appears to be the most effective, safe method for combating the loss of muscle mass, strength and functional capacity. The aim of investigators study is to develop/adopt an effective intervention specifically for elderly (65+) people with post COVID-19 condition, experiencing balance disorder and muscle weakness, in order to help them return to pre-infection mobility and function. This will be a randomized controlled study with pre- and post-intervention assessment. The participants will be recruited from nursing homes, retirement facilities, Universities of the Third Age, primary health care units (POZs), in keeping with the inclusion criteria. The patients will be randomized to one of 2 groups: RT and control (no exercise). The participants' muscle strength under dynamic condition, balance (especially fall risk), body composition and quality of life will be assessed pre- and post-intervention. The investigators main research outcome - safe exercise protocols and interventions - will be developed to match the needs of the elderly in the current pandemic (and post-pandemic) scenario, in order to maintain/improve the health, balance, muscle strength, cognitive function and, consequently, quality of life of older adults affected by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* positive Polymerase Chain Reaction test
* positive result in test for antibodies against the Severe Acute Respiratory Syndrome-Corona Virus -2 coronavirus 3-12 months prior to the study start

Exclusion Criteria:

* cardiac dysfunction,
* stress disorder,
* oxygen desaturation,
* dysfunction of the autonomic nervous system (orthostatic intolerance)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength under dynamic conditions first | Day 1
  Muscle strength will be measured under dynamic (for the knee muscles) and static conditions (for the elbow, knee, hip and ankle muscles). Both legs and arms will be tested. Isokinetic knee strength will be examined using the Biodex System 3 Professional dynamometer (Biodex Medical Systems, New York,USA) Maximal muscle strength will be defined as the highest peak torque (Newton-meters, Nm). To allow adaptation prior to the examination, subjects will be allowed to practice the motions 3 times prior to testing. Maximal Voluntary Contraction (MVC) will be measured in sitting position using 'JBA Staniak' equipment. Ankle, knee, hip and elbow joint will be standing in 90 degrees positions and isometric contraction will be calculated.The procedure will be repeated twice and isometric contraction will be held for 3 seconds in each muscle group.
Muscle strength under dynamic conditions second | Day 1
  The peak torques at angular velocities of 60°/s (5 times) and 180°/s (10 times) will be measured. To allow adaptation prior to the examination, subjects will be allowed to practice the motions 3 times prior to testing. Ankle, knee, hip and elbow joint will be standing in 90 degrees positions and isometric contraction will be calculated.The procedure will be repeated twice and isometric contraction will be held for 3 seconds in each muscle group.
Balance assessment first | Day 1
  Three protocols are prepared on the Biodex Balance System Standard Definition platform from Biodex (BBS). Each of them lasts 20 seconds. The BBS enables subjects to be tested on a stable or unstable platform on 12 levels, with the degree of instability of the platform increasing from 12 to 1 (the most stable platform being level 12).
Balance assessment second | Day 1
  The Fall Risk Test is also carried out with EO on an unstable platform at levels ranging from 12 to 8, and 6 to 2. On this basis, the fall risk index (FRI) will be determined.
Balance assessment third | Day 1
  Postural Stability Test (PST) is performed on a stationary platform with eyes open (EO) and closed (EC) to determine: an OSI (overall stability index), APSI (anterior-posterior stability index) and MLSI (medial-lateral stability index).
Balance assessment fourth | Day 1
  OSI (overall stability index)
Balance assessment fifth | Day 1
  APSI (anterior-posterior stability index)
Balance assessment sixth | Day 1
  MLSI (medial-lateral stability index).
Body Composition BMI (kg/m^2) measured by DXA (dual-energy X-ray absorptiometry) | Day 1
  During each series of testing, body composition called BMI (kg/m^2) will be evaluated using the DXA (dual-energy X-ray absorptiometry) method (GE Lunar Prodigy, GE Healthcare, Madison, Wisconsin, USA) in all participants.
Body Height BSM170 (InBody, 'Biospace Company', Japan) | Day 1
  During each series of testing, body height will be measured to the nearest 0.1 cm with digital stationmaster
Body Mass (InBody 720, 'Biospace Company', Japan) | Day 1
  During each series of testing, body mass will be determined to the nearest 0.1 kg with a medical scale

SECONDARY OUTCOMES:
Quality of life tests World Health Organization Quality of Life Scale(WHOQOL-Bref) | Day 1
  WHOQOL-Bref is a research tool used to assess quality of life in healthy and ill individuals, both for medicinal and cognitive purposes. It allows to obtain a life quality profile in the following domains: physical health, psychological health, social relationships, and environment. The scores reflect individual perceptions of life quality in these areas. Score is measured from 0 to 100 where 0 is the worst and 100 is the best result.

CONTACTS AND LOCATIONS:
Locations (1):
- AWF Warszawa, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No